CLINICAL TRIAL: NCT02127671
Title: Comprehensive Cardiovascular Diseases (CVD) Risk Reduction Trial in Persons With Serious Mental Illness
Brief Title: Intervention Trial to Decrease Cardiovascular Risk in Persons With Serious Mental Illness
Acronym: IDEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NA_00072197; R01HL112299 (NIH)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Risk Factors; Serious Mental Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDEAL intervention (Experimental): Individual cardiovascular risk reduction counseling, coordination with primary care providers to ensure appropriate management of risk factors, and collaboration with mental health staff and social supports. All participants will be offered group exercise classes, and programs will be provided with instruction to provide more healthy meals.
  Interventions: Other: IDEAL intervention
- Control (Other): All participants will be offered group exercise classes, and programs will be provided with instruction to provide more healthy meals.
  Interventions: Other: Control

INTERVENTIONS:
Other: IDEAL intervention
  Arms: IDEAL intervention
Other: Control
  Arms: Control

SUMMARY:
This study will determine whether a program where a health coach works with participants on heart healthy behaviors and treatment of risk factors is coordinated with primary care can reduce overall heart disease risk in people with serious mental illness.

DETAILED DESCRIPTION:
The objective of this study is to perform a randomized clinical trial (IDEAL) to test a comprehensive cardiovascular risk reduction program for persons with serious mental illness. This trial will enroll adult mental health consumers with at least one cardiovascular risk factor and randomize them to the 18-month IDEAL intervention or control. Intervention participants will receive individual cardiovascular risk reduction counseling, coordination with primary care providers to ensure appropriate management of risk factors, and collaboration with mental health staff and social supports to encourage and motivate participants to reach goals. All participants will be offered group exercise classes, and programs will be provided with instruction to provide more healthy meals. The primary outcome will be the change in estimated cardiovascular risk from the global Framingham Risk Score.

ELIGIBILITY:
Inclusion Criteria:

* ▪ Age 18 and older

  ▪ Body mass index at least 25 kg/m2 OR one of the following CVD risk factors:
* Hypertension (SBP>= 140mmHg or DBP>= 90mmHg or on antihypertensive medications;
* Diabetes mellitus (fasting blood sugar> 125mg/dl or hemoglobin A1c>6.5 or on a hypoglycemic medication);
* Dyslipidemia (LDL >130 mg/dl , HDL<40 or total cholesterol >=200 or on a lipid lowering agent);
* Current tobacco smoker

  * Able and willing to give informed consent
  * Completion of baseline data collection
  * Willing to accept randomization
  * Willing to participate in the intervention

Exclusion Criteria:

* ▪ Cardiovascular event (unstable angina, myocardial infarction) within the past 6 months

  * Serious medical condition which either limits life expectancy or requires active management (e.g., certain cancers)
  * Condition which interferes with outcome measurement (e.g., dialysis)
  * Pregnant or planning a pregnancy during study period. Nursing mothers would need approval from physician.
  * Alcohol or substance use disorder if not sober/abstinent for 30 days
  * Planning to leave rehabilitation center or clinic within 6 months or move out of geographic area within 18 months
  * Investigator judgment (e.g., for concerns about participant or staff safety)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2013-12-12; Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail L. Daumit, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ProHealth Clinical Research Facility, Woodlawn, Maryland, United States

REFERENCES:
- [Derived] Daumit GL, Dalcin AT, Dickerson FB, Miller ER, Evins AE, Cather C, Jerome GJ, Young DR, Charleston JB, Gennusa JV 3rd, Goldsholl S, Cook C, Heller A, McGinty EE, Crum RM, Appel LJ, Wang NY. Effect of a Comprehensive Cardiovascular Risk Reduction Intervention in Persons With Serious Mental Illness: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e207247. doi: 10.1001/jamanetworkopen.2020.7247. PMID 32530472

RESULTS

PARTICIPANT FLOW:
Groups:
- IDEAL Intervention: Individual cardiovascular risk reduction counseling, coordination with primary care providers to ensure appropriate management of risk factors, and collaboration with mental health staff and social supports. All participants will be offered group exercise classes, and programs will be provided with instruction to provide more healthy meals.
  IDEAL intervention
- Control: All participants will be offered group exercise classes, and programs will be provided with instruction to provide more healthy meals.
  Control
Period: Overall Study
Arm/Group | IDEAL Intervention | Control
Started | 132 | 137
Completed | 124 | 132
Not Completed | 8 | 5
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 4 | 2
Not completed — Physician Decision | 1 | 0
Not completed — incarceration | 0 | 1
Not completed — Did not have full Framingham risk score measured | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDEAL Intervention | Control | Total
Number analyzed (Participants) | 132 | 137 | 269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 128 | 124 | 252
  >=65 years | 4 | 13 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 71 | 141
  Male | 62 | 66 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 130 | 133 | 263
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 61 | 63 | 124
  White | 67 | 68 | 135
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 132 | 137 | 269
primary psychiatric diagnosis [Count of Participants; unit: Participants]
  schizophrenia | 40 | 41 | 81
  schizoaffective disorder | 46 | 32 | 78
  bipolar disorder | 25 | 42 | 67
  major depressive disorder | 20 | 18 | 38
  other psychotic disorder | 1 | 4 | 5
Number of cardiovascular disease (CVD) risk factors [Count of Participants; unit: Participants]
  1 cvd risk factors | 14 | 20 | 34
  2 cvd risk factors | 37 | 23 | 60
  3 cvd risk factors | 39 | 47 | 86
  4 cvd risk factors | 33 | 34 | 67
  5 cvd risk factors | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Global Framingham Risk Score
Description: Global Framingham Cardiovascular disease Risk Score. Higher score indicates higher cardiovascular risk. The score can range from 0-38 with higher scores yielding increased 10-year probability of stroke
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
score on a scale
  Baseline | 11.5 (11.5) | 12.7 (12.7)
  18 months | 9.9 (10.2) | 12.3 (12.0)
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; Test type: Superiority; Mean Difference (Net) = -12.7, 95% CI 2-sided [-22.9 to -2.5]

2. Secondary Outcome: Weight in Pounds
Description: Weight measured in pounds.
Time Frame: Baseline, 6 and 18 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
pounds
  Baseline | 219.5 (53.3) | 208.6 (48.0)
  6 month | 216.9 (49.1) | 208.3 (49.9)
  18 month | 213.2 (51.6) | 202.9 (46.9)

3. Secondary Outcome: Body Mass Index (BMI)
Description: Body mass index measured in kg/meter2
Time Frame: baseline and 18 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
kg/m^2
  Baseline | 34.4 (7.8) | 32.9 (6.6)
  18 months | 33.7 (7.7) | 32.1 (6.6)
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; Test type: Superiority; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.7 to 0.9]

4. Secondary Outcome: Distance Traveled in the 6 Minute Walk Test
Description: 6 minute walk test measured in feet. More feet traveled indicates better results.
Time Frame: Baseline, 6 and 18 months
Population: Data reported on all clients who completed measure at timepoint. Data was not modeled.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 134
feet
  Baseline | 909.5 (233.4) | 910.7 (249.6)
  6 months: number analyzed (Participants) | 110 | 105
  6 months | 922.9 (248.2) | 926.9 (239.4)
  18 months: number analyzed (Participants) | 95 | 93
  18 months | 925.1 (217.3) | 910.7 (249.6)

5. Secondary Outcome: Healthy Diet as Indicated by Sugar Sweetened Beverage Consumption
Description: Self reported number of sugar sweetened beverages consumed per week on average. A higher score indicated a greater number of sugar sweetened beverages consumed.
Time Frame: Baseline, 6 and 18 months
Population: Data reported on all clients with data collected at timepoints Data was not modeled.
Measure: Mean (Standard Deviation); unit: Sugar sweetened beverages per week
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
Sugar sweetened beverages per week
  Baseline | 8.8 (9.7) | 9.8 (9.8)
  6 month: number analyzed (Participants) | 121 | 124
  6 month | 8.4 (9.8) | 11.1 (12.9)
  18 month: number analyzed (Participants) | 115 | 119
  18 month | 9.1 (11.7) | 11.3 (12.6)

6. Secondary Outcome: Healthy Diet as Indicated by Fast Food Consumption
Description: Self reported number of times eating at a fast food restaurant per month on average. A higher score indicates a greater frequency of eating fast food.
Time Frame: baseline, 6 and 18 months
Population: Data reported on all clients with data collected at timepoints. Data was not modeled.
Measure: Mean (Standard Deviation); unit: Fast food per month
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
Fast food per month
  Baseline | 4.3 (6.5) | 3.9 (7.0)
  6 month: number analyzed (Participants) | 121 | 124
  6 month | 3.7 (5.8) | 5.2 (10.4)
  18 month: number analyzed (Participants) | 115 | 119
  18 month | 3.8 (8.5) | 3.8 (9.3)

7. Secondary Outcome: Fasting Glucose Level
Description: Fasting glucose level reported in mg/dl.
Time Frame: baseline and 18 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
mg/dl
  baseline | 106.5 (36.7) | 110.6 (36.9)
  18 months | 106.7 (45.2) | 117.4 (60.0)
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; Test type: Superiority; Mean Difference (Net) = -7.6, 95% CI 2-sided [-17.6 to 2.4]

8. Secondary Outcome: Participants With Diabetes Mellitus Treated to Goal (HgBA1c)
Description: A1c Goal used for analysis was <7.
Time Frame: Baseline, 6 and 18 months
Population: Only those with diabetes at baseline were included in analysis and data is reported on all clients with data collected at timepoints. Data was not modeled.
Measure: Count of Participants; unit: Participants
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 42 | 51
Participants
  baseline: Yes | 27 | 25
  baseline: No | 15 | 26
  6 month: number analyzed (Participants) | 41 | 47
  6 month: Yes | 29 | 23
  6 month: No | 12 | 24
  18 month: number analyzed (Participants) | 38 | 48
  18 month: Yes | 31 | 26
  18 month: No | 7 | 22
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.3 to 0.2]

9. Secondary Outcome: Current Smoking Status
Description: Self reported smoking status for clients with the data below reflecting the number of clients who reported currently smoking at that time point.
Time Frame: Baseline and 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
Participants
  Baseline | 65 | 73
  18 months | 47 | 67
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; Test type: Superiority; Mean Difference (Net) = -10.5, 95% CI 2-sided [-18.4 to -2.6]

10. Secondary Outcome: Blood Pressure
Description: Systolic and diastolic blood pressure measured in mmhg
Time Frame: baseline and 18 months
Measure: Mean (Standard Deviation); unit: mmhg
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
mmhg
  Baseline systolic blood pressure | 118.0 (13.0) | 116.5 (12.9)
  Baseline diastolic blood pressure | 75.3 (8.2) | 74.9 (9.3)
  18 month systolic blood pressure | 120.1 (14.5) | 120.2 (16.2)
  18 month diastolic blood pressure | 73.9 (9.2) | 74.7 (11.1)
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; systolic; Test type: Superiority; Mean Difference (Net) = -1.8, 95% CI 2-sided [-5.1 to 1.5]
Statistical Analysis 2: Comparison: IDEAL Intervention vs Control; diastolic; Test type: Superiority; Mean Difference (Net) = -1.7, 95% CI 2-sided [-3.8 to 0.5]

11. Secondary Outcome: Participants With Hypertension Treated to Goal
Description: Hypertension goal used for analysis was systolic blood pressure <140 and diastolic blood pressure <90. not modeled
Time Frame: Baseline, 6 and 18 months
Population: Only those with hypertension at baseline were included in analysis and data is reported on all clients with data collected at timepoints. Data was not modeled.
Measure: Count of Participants; unit: Participants
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 72 | 70
Participants
  baseline: Yes | 61 | 54
  baseline: No | 11 | 16
  6 month: number analyzed (Participants) | 70 | 68
  6 month: Yes | 62 | 55
  6 month: No | 8 | 13
  18 months: number analyzed (Participants) | 65 | 68
  18 months: Yes | 57 | 51
  18 months: No | 8 | 17

12. Secondary Outcome: Total Cholesterol
Description: Total cholesterol measured in mg/dl
Time Frame: Baseline and 18 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
mg/dl
  baseline | 178.9 (42.1) | 181.1 (41.6)
  18 month | 171.8 (38.3) | 177.7 (48.7)
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; Test type: Superiority; Mean Difference (Net) = -4.3, 95% CI 2-sided [-13.3 to 4.7]

13. Secondary Outcome: LDL Cholesterol
Description: LDL cholesterol measured in mg/dl
Time Frame: Baseline and 18 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
mg/dl
  baseline | 101.9 (36.8) | 101.0 (33.4)
  18 months | 93.7 (33.5) | 97.3 (35.9)
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; Test type: Superiority; Mean Difference (Net) = -5.4, 95% CI 2-sided [-12.7 to 2.0]

14. Secondary Outcome: HDL Cholesterol
Description: HDL cholesterol measured in mg/dl
Time Frame: Baseline and 18 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
mg/dl
  baseline | 49.2 (15.3) | 50.2 (19.3)
  18 months | 50.7 (14.8) | 51.0 (17.7)
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; Test type: Superiority; Mean Difference (Net) = 1.0, 95% CI 2-sided [-1.8 to 3.8]

15. Secondary Outcome: Triglycerides
Description: Triglycerides measured in mg/dl
Time Frame: Baseline and 18 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
mg/dl
  baseline | 140.2 (74.3) | 156.6 (106.7)
  18 months | 141.0 (76.9) | 149.0 (111.1)
Statistical Analysis 1: Comparison: IDEAL Intervention vs Control; Test type: Superiority; Mean Difference (Net) = 8.1, 95% CI 2-sided [-13.4 to 29.6]

16. Secondary Outcome: Participants With Dyslipidemia Treated to Goal
Description: Goal used for analysis was LDL cholesterol < 130 mg/dl and Total cholesterol < 200mg/dl.
Time Frame: Baseline, 6 and 18 months
Population: Only those with dyslipidemia at baseline were included in analysis and data is reported on all clients with data collected at timepoints. Data was not modeled.
Measure: Count of Participants; unit: Participants
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 82 | 93
Participants
  Baseline: Yes | 46 | 53
  Baseline: No | 36 | 40
  6 month: number analyzed (Participants) | 76 | 84
  6 month: Yes | 47 | 55
  6 month: No | 29 | 29
  18 month: number analyzed (Participants) | 75 | 87
  18 month: Yes | 57 | 63
  18 month: No | 18 | 24

17. Other Pre Specified Outcome: Health Status With Short Form (SF)-12
Description: Health status reported for the SF-12 in two subscales-physical component summary (PCS) and the mental component summary (MCS). Both subscale score ranges are 0-100. Higher scores indicate better physical or mental health.
Time Frame: Baseline, 6 and 18 months
Population: Participants with data collected at the timepoints
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
score on a scale
  Physical - Baseline | 45.3 (9.1) | 43.9 (10.0)
  Physical - 6 months: number analyzed (Participants) | 120 | 122
  Physical - 6 months | 45.2 (9.3) | 44.0 (9.1)
  Physical - 18 months: number analyzed (Participants) | 113 | 120
  Physical - 18 months | 46.8 (8.4) | 44.6 (8.9)
  Mental - Baseline | 47.3 (8.3) | 47.9 (8.5)
  Mental - 6 months: number analyzed (Participants) | 120 | 122
  Mental - 6 months | 48.7 (8.1) | 48.2 (7.2)
  Mental - 18 months: number analyzed (Participants) | 113 | 120
  Mental - 18 months | 49.3 (7.7) | 48.7 (8.3)

18. Other Pre Specified Outcome: Quality of Life Based on the EUROQOL
Description: Self reported measured by the EUROQOL EQ-5D-3L. A higher score indicates better health and a lower score indicates worse health; on a scale of 0 to 1. Not modeled.
Time Frame: Baseline, 6 and 18 months
Population: Data reported on all clients with data collected at timepoints. Data was not modeled.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
score on a scale
  Baseline | 0.75 (0.20) | 0.74 (0.20)
  6 months: number analyzed (Participants) | 120 | 122
  6 months | 0.77 (0.20) | 0.76 (0.19)
  18 months: number analyzed (Participants) | 114 | 120
  18 months | 0.82 (0.19) | 0.79 (0.20)

19. Other Pre Specified Outcome: Medication Adherence
Description: Used medication adherence measure designed by Morisky et al and separately evaluated somatic and psychiatric medications.
Time Frame: Baseline, 6 and 18 months
Population: Data reported on all clients with data collected at timepoints. Data was not modeled.
Measure: Count of Participants; unit: Participants
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
Participants
  Somatic - Baseline: Good adherence | 45 | 51
  Somatic - Baseline: Moderate adherence | 39 | 41
  Somatic - Baseline: Poor adherence | 21 | 26
  Somatic - Baseline: Reported not taking medication type | 27 | 19
  Somatic - 6 months: number analyzed (Participants) | 122 | 125
  Somatic - 6 months: Good adherence | 39 | 45
  Somatic - 6 months: Moderate adherence | 43 | 41
  Somatic - 6 months: Poor adherence | 28 | 25
  Somatic - 6 months: Reported not taking medication type | 12 | 14
  Somatic - 18 months: number analyzed (Participants) | 115 | 121
  Somatic - 18 months: Good adherence | 49 | 46
  Somatic - 18 months: Moderate adherence | 31 | 43
  Somatic - 18 months: Poor adherence | 23 | 22
  Somatic - 18 months: Reported not taking medication type | 12 | 10
  Psychiatric - Baseline: Good adherence | 40 | 49
  Psychiatric - Baseline: Moderate adherence | 54 | 50
  Psychiatric - Baseline: Poor adherence | 37 | 37
  Psychiatric - Baseline: Reported not taking medication type | 1 | 1
  Psychiatric - 6 months: number analyzed (Participants) | 122 | 125
  Psychiatric - 6 months: Good adherence | 33 | 43
  Psychiatric - 6 months: Moderate adherence | 50 | 42
  Psychiatric - 6 months: Poor adherence | 38 | 39
  Psychiatric - 6 months: Reported not taking medication type | 1 | 1
  Psychiatric - 18 months: number analyzed (Participants) | 115 | 121
  Psychiatric - 18 months: Good adherence | 41 | 41
  Psychiatric - 18 months: Moderate adherence | 49 | 40
  Psychiatric - 18 months: Poor adherence | 25 | 38
  Psychiatric - 18 months: Reported not taking medication type | 0 | 2

20. Other Pre Specified Outcome: Medication Use for Cardiovascular Risk Factors
Description: Medications as reported by participant and then categorized by research study nurse into hypertension, diabetes, dyslipidemia and smoking cessation. Will report the number of participants taking at least one medication in each category of those with the specified condition at baseline.
Time Frame: Baseline, 6 and 18 months
Population: Only includes those with specified condition at baseline were included in analysis and data is reported on all clients with data collected at timepoints. Data was not modeled.
Measure: Count of Participants; unit: Participants
Arm/Group | IDEAL Intervention | Control
Number analyzed (Participants) | 132 | 137
Participants
  Hypertension - Baseline: number analyzed (Participants) | 72 | 70
  Hypertension - Baseline: Reported medication for risk factor | 6 | 5
  Hypertension - Baseline: Did not report medication for risk factor | 66 | 65
  Hypertension - 6 months: number analyzed (Participants) | 68 | 67
  Hypertension - 6 months: Reported medication for risk factor | 59 | 55
  Hypertension - 6 months: Did not report medication for risk factor | 9 | 12
  Hypertension - 18 months: number analyzed (Participants) | 58 | 58
  Hypertension - 18 months: Reported medication for risk factor | 51 | 47
  Hypertension - 18 months: Did not report medication for risk factor | 7 | 11
  Diabetes - Baseline: number analyzed (Participants) | 42 | 51
  Diabetes - Baseline: Reported medication for risk factor | 33 | 41
  Diabetes - Baseline: Did not report medication for risk factor | 9 | 10
  Diabetes - 6 months: number analyzed (Participants) | 39 | 47
  Diabetes - 6 months: Reported medication for risk factor | 35 | 41
  Diabetes - 6 months: Did not report medication for risk factor | 4 | 6
  Diabetes - 18 months: number analyzed (Participants) | 34 | 41
  Diabetes - 18 months: Reported medication for risk factor | 29 | 37
  Diabetes - 18 months: Did not report medication for risk factor | 5 | 4
  Dyslipidemia - Baseline: number analyzed (Participants) | 82 | 92
  Dyslipidemia - Baseline: Reported medication for risk factor | 59 | 75
  Dyslipidemia - Baseline: Did not report medication for risk factor | 23 | 17
  Dyslipidemia - 6 months: number analyzed (Participants) | 77 | 85
  Dyslipidemia - 6 months: Reported medication for risk factor | 54 | 68
  Dyslipidemia - 6 months: Did not report medication for risk factor | 23 | 17
  Dyslipidemia - 18 months: number analyzed (Participants) | 69 | 79
  Dyslipidemia - 18 months: Reported medication for risk factor | 49 | 61
  Dyslipidemia - 18 months: Did not report medication for risk factor | 20 | 18
  Smoking cessation - Baseline: number analyzed (Participants) | 65 | 72
  Smoking cessation - Baseline: Reported medication for risk factor | 6 | 1
  Smoking cessation - Baseline: Did not report medication for risk factor | 59 | 71
  Smoking cessation - 6 months: number analyzed (Participants) | 60 | 67
  Smoking cessation - 6 months: Reported medication for risk factor | 12 | 3
  Smoking cessation - 6 months: Did not report medication for risk factor | 48 | 64
  Smoking cessation - 18 months: number analyzed (Participants) | 55 | 60
  Smoking cessation - 18 months: Reported medication for risk factor | 14 | 3
  Smoking cessation - 18 months: Did not report medication for risk factor | 41 | 57

ADVERSE EVENTS:
Time Frame: baseline to 18 months
Arm/Group | IDEAL Intervention | Control
All-Cause Mortality (participants affected / at risk) | 2/132 | 2/137
Serious Adverse Events (participants affected / at risk) | 29/132 | 35/137
Other Adverse Events (participants affected / at risk) | 0/132 | 0/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDEAL Intervention (N=132) | Control (N=137)
psychiatric hospitalization (Psychiatric disorders) | 10 (14) | 9 (13)
medical hospitalization (General disorders) | 20 (22) | 30 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT02127671/Prot_SAP_000.pdf